CLINICAL TRIAL: NCT00529659
Title: A Phase IIa Randomized, Placebo-Controlled Clinical Trial to Study the Efficacy and Safety of MK-0773 in Patients With Sarcopenia
Brief Title: A Study of the Safety and Efficacy of MK-0773 in Women With Sarcopenia (Loss of Muscle Mass)(MK-0773-005)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0773-005; 2007_532
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Results first posted 2012-07-02 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-01

CONDITIONS: Sarcopenia
Keywords: Sarcopenia (loss of muscle mass)
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MK-0773 (Experimental): MK-0773
  Interventions: Drug: Comparator: MK-0773
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Comparator: MK-0773 — MK-0773 50 mg tablets twice daily, 6 month treatment period
  Arms: MK-0773
Drug: Comparator: Placebo — Placebo tablets twice daily, 6 month treatment period
  Arms: Placebo

SUMMARY:
A study to evaluate the safety, tolerability, and efficacy of MK-0773 in women with sarcopenia (loss of muscle mass).

ELIGIBILITY:
Inclusion Criteria:

* Patient is a woman who is 65 years of age or older
* Patient's lean body mass is at least 1 standard deviation below the mean of a healthy young adult population
* Patient has difficulty climbing 10 steps or walking outside on level ground for 1/4 mile without resting or Activity Measure for Post Acute Care (AM-PAC)<66

Exclusion Criteria:

* Patient has serious neurological, rheumatologic, cardiac, respiratory, kidney, psychiatric conditions
* Patient has a history of certain types of cancer

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 170 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Papanicolaou DA, Ather SN, Zhu H, Zhou Y, Lutkiewicz J, Scott BB, Chandler J. A phase IIA randomized, placebo-controlled clinical trial to study the efficacy and safety of the selective androgen receptor modulator (SARM), MK-0773 in female participants with sarcopenia. J Nutr Health Aging. 2013;17(6):533-43. doi: 10.1007/s12603-013-0335-x. PMID 23732550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized from 28 sites (2 sites in Mexico, 10 sites in South America, 8 sites in Europe, 5 sites in Asia Pacific, and 3 sites in South Africa).
Pre-assignment Details: After a 2-week placebo run-in period, patients were randomized in a 1:1 ratio to receive treatment with either oral MK-0773 50 mg twice daily or matching placebo.
Groups:
- MK-0773: MK-0773 was administered orally twice daily (BID) at a dose of 50 mg.
- Placebo: Placebo administered orally twice daily.
Period: Overall Study
Arm/Group | MK-0773 | Placebo
Started | 81 | 89
Completed | 70 | 66
Not Completed | 11 | 23
Not completed — Adverse Event | 8 | 7
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 2 | 6
Not completed — Withdrawal by Subject | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0773 | Placebo | Total
Number analyzed (Participants) | 81 | 89 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.0 (6.7) | 76.8 (7.1) | 75.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 89 | 170
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Participant Lean Body Mass
Time Frame: Baseline, Month 6
Population: The full analysis set (FAS) included all participants that received at least one dose of the study therapy and had a post-randomization measurement of lean body mass.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | MK-0773 | Placebo
Number analyzed (Participants) | 65 | 60
kg | 1.26 (1.09) | 0.29 (1.29)

2. Secondary Outcome: Change From Baseline in Participant Short Physical Performance Battery (SPPB)
Description: The Short Physical Performance Battery (SPPB) is an objective assessment tool for evaluating lower extremity functioning in older persons. The SPPB consists of 3 types of physical maneuvers: balance test, speed gait test, and chair stand test. Results from each maneuvers test are scored on a scale of 0 to 4, with an increasing composite score indicating an improved function level. The total maximum score of SPPB is 12.
Time Frame: Baseline, Month 6
Population: N = Number of participants with at least one non-missing measurement at the time point.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-0773 | Placebo
Number analyzed (Participants) | 66 | 63
Score on a Scale | 0.92 (1.63) | 0.88 (1.60)

3. Primary Outcome: Change From Baseline in Bilateral Leg Press (BLP) Measurement
Description: BLP measurements were obtained with the participant sitting on the BLP exercise machine with flexed hips and knees. The participant held the handgrips with hips flexion and knees bent at a 90 degree angle and feet placed evenly on the footpad with heels placed approximately shoulder width apart. Participants were asked to slowly push the footpad forward, while keeping the knees slightly flexed, and bend back again slowly for one repetition. The BLP procedure measures the maximum amount of weight that the patient can push through his or her full range of motion one time.
Time Frame: Baseline, Month 6
Population: N = Number of participants with at least one non-missing measurement at the time point.
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | MK-0773 | Placebo
Number analyzed (Participants) | 66 | 63
lbs | 17.42 (26.04) | 15.95 (27.84)

4. Secondary Outcome: Change From Baseline in Participant Gait Speed
Time Frame: Baseline, Month 6
Population: N = Number of participants with at least one non-missing measurement at the time point.
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | MK-0773 | Placebo
Number analyzed (Participants) | 66 | 63
cm/sec | 6.24 (17.65) | 8.91 (15.05)

5. Secondary Outcome: Change From Baseline in Stair Climbing Power
Description: Stair-climbing power is an alternate measure of lower extremity muscle strength. Participants were asked to climb a standardized 4-step flight of stairs. The study coordinator timed how long it took the participant to walk up the stairs as quickly as possible. The test starts when the tester says "go" and ends when both of the patient's feet are flat on the platform area at the top of the staircase. Participants were permitted to use the railing, and/or an assistive device, if needed. Stair climbing power was calculated as = participant weight × gravity constant × height of stairs / time.
Time Frame: Baseline, Month 6
Population: The FAS included all participants that received at least one dose of the study therapy and had a post-randomization stair climbing power measurement.
Measure: Mean (Standard Deviation); unit: watts
Arm/Group | MK-0773 | Placebo
Number analyzed (Participants) | 65 | 63
watts | 19.68 (23.85) | 14.98 (20.71)

6. Secondary Outcome: Change From Baseline in Activity Measure for Post Acute Care (AM-PAC) Physical Movement Score
Description: The Activity Measure for Post Acute Care (AM-PAC) measures function in three domains: basic mobility, daily activities, and applied cognitive function. AM-PAC scores in each functional domain have a mean of 50 with a standard deviation of 10 and scores are distributed along a continuum of function. The AM-PAC tracks outcomes as a participant progresses across an episode of care with higher scores indicating an improved level of functioning.
Time Frame: Baseline, Month 6
Population: N = Number of patient with at least one non-missing measurement at the time point.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | MK-0773 | Placebo
Number analyzed (Participants) | 65 | 63
Score on a Scale
  Baseline | 59.79 (6.29) | 59.13 (5.28)
  Change from Baseline | 2.52 (4.98) | 2.38 (4.55)

ADVERSE EVENTS:
Arm/Group | MK-0773 | Placebo
Serious Adverse Events (participants affected / at risk) | 12/81 | 9/89
Other Adverse Events (participants affected / at risk) | 50/81 | 52/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0773 (N=81) | Placebo (N=89)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distention (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medical device complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0773 (N=81) | Placebo (N=89)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Subendocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Addison's disease (Endocrine disorders) | 1 (1) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (General disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 6 (6) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medical device complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (8) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 1 (1)
Blood cortisol decreased (Investigations) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Haematocrit increased (Investigations) | 8 (8) | 2 (2)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 3 (3) | 1 (1)
High density lipoprotein decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal carcinoma (Nervous system disorders) | 2 (2) | 1 (1)
Dysstasia (Nervous system disorders) | 0 (0) | 1 (1)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Varicose ulceration (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days